CLINICAL TRIAL: NCT05148286
Title: Albumin and Crystalloid Administration in Septic Shock (ALCAMIST): Multi-center, Open Labelled Randomized Controlled Trial
Brief Title: Albumin and Crystalloid Administration in Septic Shock
Acronym: ALCAMIST
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Samsung Medical Center (Other); Gangnam Severance Hospital (Other); Chungnam National University Hospital (Other); Seoul National University Hospital (Other); Seoul National University Bundang Hospital (Other); SMG-SNU Boramae Medical Center (Other); Hanyang University (Other); Korea University Ansan Hospital (Other)
Responsible Party: Principal Investigator, Won Young Kim, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALCAMIST trial
Record Dates: First submitted 2021-11-25; First posted 2021-12-08 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Septic Shock
Keywords: Septic shock; Fluid resuscitation; Albumin; Crystalloid
MeSH Terms: conditions — Shock, Septic | interventions — Therapeutics; Albumins; Crystalloid Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): For the treatment group, 200cc of 20% human albumin with 15 cc per kg of crystalloid will be administered over 1~2h for initial fluid resuscitation.
  Interventions: Drug: Treatment
- Control (Placebo Comparator): For the control group, 30 cc per kg of crystalloid will be administered according to the usual practice.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Treatment — For the treatment group, 200cc of 20% human albumin with 15 cc per kg of crystalloid will be administered over 1~2h for initial fluid resuscitation. The treating physicians can choose the type of fluid, such as balanced fluid or isotonic saline.
  Other Names: Albumin and crystalloid
  Arms: Treatment
Drug: Placebo — For the control group, 30 cc per kg of crystalloid will be administered according to the usual practice. The treating physicians can choose the type of fluid, such as balanced fluid or isotonic saline.
  Other Names: Crystalloid only
  Arms: Control

SUMMARY:
The current guideline emphasizes fluid resuscitation as the mainstay of initial management for septic shock. Albumin has the oncotic activity to maintain intravascular volumes with additional beneficial properties in sepsis. Prior studies showed that the replacement of albumin might have survival advantages in patients with septic shock. The investigators aim to assess whether the early administration of albumin with crystalloid as initial fluid resuscitation improves survival in patients with septic shock compared to resuscitation without albumin.

DETAILED DESCRIPTION:
Sepsis is a leading cause of mortality worldwide, contributing to an estimated 11 million deaths in 2017-or 20% of all global deaths. Due to recent advances in the medical management and treatment of sepsis, the mortality of sepsis has been declined in these years, but still stayed at a high level. From 2004, the Surviving Sepsis Campaign (SSC) suggested a protocolized bundle therapy to facilitate implementation at the bedside with a defined target. Recent guideline states that this resuscitation bundle treatment should be initiated within 1 h of the emergency department (ED) triage time, named as 1-h bundle.

Fluid resuscitation, which is the mainstay of treatment to restore a patient's tissue perfusion, is associated with outcome in emergency department patients. The current guideline recommends that crystalloid for initial fluid resuscitation in sepsis and albumin can be additionally administered when patients require substantial amounts of crystalloid. Besides its oncotic functions to provide adequate intravascular volume, albumin has several beneficial properties for sepsis patients, including binding and transport of various endogenous molecules, anti-inflammatory and anti-oxidative effects, and modulation of nitric oxide metabolism. In 2004, a large randomized, prospective, double-blind study was performed in 7000 critically ill patients (SAFE study) to evaluate the effect of volume replacement therapy with human albumin on the outcome compared to only crystalloid. Although the survival rates were similar between the groups, a post hoc analysis of 1218 patients with severe sepsis showed improved survival in the albumin group compared to crystalloid alone. Furthermore, the ALBumin Italian Outcome Sepsis (ALBIOS) study investigated the effect of albumin administration and maintenance of serum albumin concentrations to at least 30 g/l on outcome in patients with severe sepsis and septic shock. This study showed a similar result to SAFE study that no difference on the outcome between the groups. Nevertheless, in the 1121 patients with septic shock, 90-day mortality was lower in the albumin group (564 patients) than in the non-albumin group (43.6 vs. 49%, p = 0.03). Recently, a retrospective study which evaluated the effect of administration of albumin combined with crystalloids in septic patients showed improved survival in 28 days. Therefore, accumulating evidence suggests that early albumin administration may provide a survival benefit in patients with severe and advanced sepsis. However, no prospective, randomized trial has adequately studied this hypothesis in patients with septic shock.

The aim of the ALCAMIST (ALbumin and Crystalloid AdMinistration In SepTic shock) study is to investigate the effect of albumin and crystalloid administration as an initial fluid choice in septic shock compared to crystalloid alone on patient survival.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years) who visit an ED directly and are suspected of sepsis with shock
* Shock is defined as hypotension (mean arterial blood pressure (MAP) < 65 or systolic blood pressure < 80) and tissue hypoperfusion such as an initial serum lactate level ≥ 4 mmol/dL.

Exclusion Criteria:

* patients who are transferred from another hospital after initial fluid administration
* patients who have set limitations on treatment (e.g. patients with a signed do-not-resuscitate order)
* patients with moribund conditions with life expectancy less than 28 days due to secondary diseases or advanced malignant disease and palliative situations with life expectancy less than 6 months
* patients who have been administered albumin before enrollment
* patients who have known hypersensitivity to albumin
* Clinical conditions, where albumin administration may be unfavorable (e.g. pulmonary edema, congestive heart failure, traumatic brain injury)
* lactation
* patients who do not voluntarily consent to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2426 (Estimated)
Dates: Start 2022-01-17 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
28-day all-cause mortality | 28-days
  The 28-day all-cause mortality in septic shock patient after admission will be evaluated

SECONDARY OUTCOMES:
90-day all-cause mortality | 90 days
  All-cause death within 90 days
ICU mortality | 28 days
  All-cause death during ICU admission
Hospital mortality | 28 days
  All-cause death during hospitalization
The Sequential organ Failure Assessment (SOFA) score | 28 days
  The SOFA score will be recorded daily up to 28 days after randomization. Death within 72 hours will be counted as the maximum SOFA score.
Intensive Care Unit (ICU) stay | 90 days
  The total length of ICU stay will be determined from the date of ICU admission until the patient is discharged from the ICU or the date of death from any cause, assessed up to 90 days after the first day of admission.
7-day mortality | 7 days
  All-cause death within 7 days
Ventilator free days | 28 days
  Days without ventilator within 28 days from admission
Vasopressor free days | 28 days
  Days without vasopressor within 28 days from admission
Total amount of fluid administration | 3 day, 7 day, 28 day
  Total amount of fluid administration during hospital admission
Total fluid balance | 28 days
  Fluid balance will be recorded daily up to 28 days after randomization
Maximum dose of vasopressor use | 28 days
  Maximum dose of vasopressor during hospital admission
Renal replacement therapy | 28 days
  Whether renal replacement therapy was initiated during hospital admission after randomization.
Safety-related parameters | 28 days
  Occurrence of adverse event, serious adverse event (e.g. anaphylactic shock, hypervolemia, pulmonary edema)

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No